CLINICAL TRIAL: NCT02899312
Title: Fluorine-18 - 2-(3-(1-carboxy-5-[(6-[18F]Fluoro-pyridine-3-carbonyl)-Amino]-Pentyl)-Ureido)-Pentanedioic Acid (18F-DCFPyL) Positron Emission Tomography / Computed Tomography (PET/CT) for Assessment of Recurrent Prostate Cancer
Brief Title: PSMA PET/CT for Assessment of Recurrent Prostate Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: H16-01551
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PSMA PET/CT scan — All participants will undergo the same procedures listed in "Detailed Description" in the protocol section.
  Other Names: 18F-DCFPyL PET/CT

SUMMARY:
Prostate cancer (PC) is the third most common cause of cancer death in men. Most patients with localized PC will be cured with surgery or radiation therapy, but up to 35% of patients will have their PC return. Whether it has returned locally or distantly determines which type of treatment they will receive. Current conventional imaging modalities have limitations particularly at low prostate-specific antigen (PSA) levels. This study proposes to use Fluorine-18-2-(3-(1-carboxy-5-[(6-[18F]fluoro-pyridine-3-carbonyl)-amino]-pentyl)-ureido)-pentanedioic acid (18F-DCFPyL) Positron Emission Tomography / Computer Tomography (PET/CT) scans which targets prostate-specific membrane antigens (PSMA) to detect where in the body the PC has recurred.

DETAILED DESCRIPTION:
This is a prospective single cohort study to evaluate the diagnostic utility of 18F-DCFPyL PET/CT in detecting sites of recurrent prostate cancer, in patients who have negative or equivocal findings on conventional imaging. Eligible subjects will undergo a 18F-DCFPyL PET/CT at the British Columbia Cancer Agency (BCCA) - Vancouver Centre.

18F-DCFPyL- Each subject will receive an 18F-DCFPyL PET/CT scan at the BCCA - Vancouver Centre, as part of this research study. Each study subject will receive a bolus intravenous dose of 18F-DCFPyL. The subject will rest in a comfortable chair for 120 minutes and will then be taken to the PET/CT scanner for images. The PET/CT scan will take approximately three hours extra of patient time above and beyond the time needed for standard of care.

Medical History Questionnaire- Demographic and medical history data will be collected either in person before the PET scan appointment or by mail or phone, whichever is the most convenient to the subject.

Follow-up assessments- Positive 18F-DCFPyL findings should be investigated and correlated with other imaging modalities and/or biopsy whenever possible. These additional procedures are left at the discretion of the referring physician for the clinical management of their patient, and will not be mandated by the study. The results of such investigations will be captured during the follow-up period, to verify the accuracy of 18F-DCFPyL findings.

All subjects will be requested to either return to the functional imaging department approximately 24 hours (acceptable range 16-28 hours) after the injection of 18F-DCFPyL or agree to be contacted by phone. The subjects will be asked if they experienced any undesirable effects following the administration of 18F-DCFPyL, or in the intervening 24 hours. The local site attending nuclear medicine physician will then make an assessment as to whether these effects are likely related to 18F-DCFPyL administration.

All subjects will receive up to three clinical follow-up evaluations at 12, 24 and 36 months following the 18F-DCFPyL PET/CT exam to assess the presence of recurrence, once presence of recurrence is confirmed follow-up will be discontinued. The evaluation will include a chart review of available imaging, laboratory tests, and treatment along with review of any symptoms. The data required can be obtained from a review of the patient's paper and electronic charts, supplemented by telephone contact as needed to complete the information. The treating oncologist will fill out a survey to determine the clinical impact of the 18F-DCFPyL on clinical managements. This will be categorized into 'minor' (change in treatment site or dose) or 'major' (change in treatment modality).

ELIGIBILITY:
Inclusion Criteria:

* Known PC with a biochemical recurrence (BR) after initial curative therapy with radical prostatectomy, with a documented history of failure of PSA to fall to undetectable levels (PSA persistence) or undetectable PSA after radical prostatectomy with a subsequent detectable PSA that increased on 2 or more determinations (PSA recurrence). The patient may have received treatment following documentation of PSA persistence or PSA recurrence. The most recent PSA measurement must be greater than 0.4 ng/mL.
* Participants with findings on other examinations (such as plain x-ray, CT, MRI or bone scintigraphy and others) that are suspicious for metastatic disease but not conclusively diagnostic of metastatic disease.
* Known PC with BR after initial curative therapy with radiation therapy (including brachytherapy), with a PSA level >2 ng/mL above the nadir after radiation therapy.
* Castration resistant PC with a minimum PSA of 2.0 ng/mL with 2 consecutive rises above the nadir and castrate levels of testosterone (<1.7 nmol/L). Treatment does not need to be discontinued before the 18F-DCFPyL scan.
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less.

Exclusion Criteria:

* Medically unstable (eg. acute illness, unstable vital signs)
* Unable to lie supine for the duration of imaging
* Unable to provide written consent
* Exceeds safe weight limit of the PET/CT bed (204.5 kg) or unable to fit through the PET/CT bore (diameter 70 cm)

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The purpose of this study is to evaluate the diagnostic utility of 18F-DCFPyL PET/CT in identifying sites of prostate cancer recurrence where conventional imaging has been negative or equivocal. Concordance with histology, imaging or follow up will be assessed. This study will also assess the clinical impact of 18F-DCFPyL PET/CT on patient management.
Sampling Method: Non-Probability Sample
Enrollment: 2244 (Estimated)
Dates: Start 2017-03-16 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
superiority of 18F-DCFPyL PET/CT over conventional imaging for detection of recurrent prostate cancer. | 3 years after the PSMA PET scan
  Comparison to conventional imaging studies, pathology and clinical follow-up up to 3 years after PSMA imaging.

SECONDARY OUTCOMES:
clinical impact of 18F-DCFPyL PET/CT | 6 months after the PSMA PET scan
  To assess the clinical impact of 18F-DCFPyL scans inpatient management. Eg, surgical resection or localized radiation.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Benard, MD, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available?

REFERENCES:
- [Derived] Harsini S, Martineau P, Plaha S, Saprunoff H, Chen C, Bishop J, Tyldesley S, Wilson D, Benard F. Prognostic significance of a negative PSMA PET/CT in biochemical recurrence of prostate cancer. Cancer Imaging. 2024 Aug 30;24(1):117. doi: 10.1186/s40644-024-00752-1. PMID 39210431
- [Derived] Harsini S, Wilson D, Saprunoff H, Allan H, Gleave M, Goldenberg L, Chi KN, Kim-Sing C, Tyldesley S, Benard F. Outcome of patients with biochemical recurrence of prostate cancer after PSMA PET/CT-directed radiotherapy or surgery without systemic therapy. Cancer Imaging. 2023 Mar 17;23(1):27. doi: 10.1186/s40644-023-00543-0. PMID 36932416